CLINICAL TRIAL: NCT04351672
Title: Time-restricted Feeding as a Dietary Strategy Against Metabolic Disturbances in Humans
Acronym: ChronoFast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: Charite University, Berlin, Germany (Other); Immanuel Krankenhaus Berlin, Germany (Unknown); Hasso-Plattner Institut, Potsdam, Germany (Unknown); University of Potsdam (Other)
Responsible Party: Principal Investigator, Olga Ramich (formerly Pivovarova), project director, German Institute of Human Nutrition
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DFG RA 3340/3-1
Record Dates: First submitted 2020-04-07; First posted 2020-04-17 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Overweight and Obesity
Keywords: Time-restricted feeding; Meal timing; Obesity; Glycemic control; Blood lipids; Inflammation; Sleep
MeSH Terms: conditions — Overweight; Obesity; Intermittent Fasting; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Time-Restricted Feeding (Experimental)
  Interventions: Behavioral: Early Time-Restricted Feeding
- Late Time-Restricted Feeding (Experimental)
  Interventions: Behavioral: Late Time-Restricted Feeding

INTERVENTIONS:
Behavioral: Early Time-Restricted Feeding — Eat between 8 am and 4 pm for two weeks
  Other Names: Early TRF; eTRF
  Arms: Early Time-Restricted Feeding
Behavioral: Late Time-Restricted Feeding — Eat between 1 pm and 9 pm for two weeks
  Other Names: Late TRF; lTRF
  Arms: Late Time-Restricted Feeding

SUMMARY:
This human dietary intervention study with a cross-over design aims to compare the effects of two isocaloric diets - early time-restricted feeding (TRF) vs. late TRF - on glycemic control and lipid metabolism in overweight and obese women.

DETAILED DESCRIPTION:
The participants are randomly allocated to one of two study groups: In study group (A) participants will begin with the early TRF (e-TRF) intervention. They will consume their habitual food (and the habitual daily amount of food) between 8 am and 4 pm for two weeks. After a washout-phase participants will conduct the late TRF (l-TRF) and consume their habitual food between 1 pm and 9 pm for another two weeks. Study group (B) receives the same interventions in the reversed order. Both dietary regimens will result in 8-hr eating period and 16-hr fasting period during the 24h day.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-35 kg/m²

Exclusion Criteria:

* prior diagnosis of type 1 or 2 diabetes
* weight changes > 5% within past 3 months
* current shift work or history of shift work
* traveled across more than one time zone one month before the study
* poor quality of sleep (PSQI score>10)
* eating disorders, food intolerance/allergy, severe indigestion
* Pregnant or breastfeeding
* severe internal or psychiatric disorders or other conditions that might influence the outcome of the study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 2 weeks
  Assessed using Matsuda index in oral glucose tolerance test (OGTT)

SECONDARY OUTCOMES:
Glucose tolerance, fasting glucose, and overall daily glycemic variation | 2 weeks (OGTT) and 14 days (CGM)
  Assessed by glucose area under the curve in OGTT and using a continuous glucose monitoring (CGM)
Metabolic hormones and inflammatory markers | 2 weeks
  Levels of hormones related to the glucose metabolism, hormones of appetite regulation, adipokines and inflammatory markers
Oxidative stress markers | 2 weeks
  Malondialdehyde, 3-nitrotyrosine, and protein carbonyls
Blood lipids | 2 weeks
  Total cholesterol, low-density lipoprotein and high-density lipoprotein cholesterol and triglycerides
Blood pressure | 2 weeks
  Systolic and diastolic blood pressure
Liver enzymes | 2 weeks
  γ-glutamyltransferase (GGT), aspartate aminotransferase (ALT), and alanine aminotransferase (AST)
Anthropometric parameters: body weight | 2 weeks
  Body weight in kilograms
Anthropometric parameters: BMI | 2 weeks
  BMI in kg/m^2
Anthropometric parameters: waist circumference | 2 weeks
  Waist circumference in centimeters
Anthropometric parameters: fat and lean mass | 2 weeks
  Fat and lean mass in kilograms assessed by bioelectrical impedance analysis
Food intake: eating times | 14 days
  Eating times in hours and minutes as assessed by food records
Food intake: calorie intake | 14 days
  Calorie intake in kilocalories as assessed by food records
Food intake: macronutrient composition | 14 days
  Macronutrient composition in percentage of energy intake as assessed by food records
Satiety and hunger scores | 2 weeks
  Assessed using Visual Analog Scales (VAS with a scale of 1-100, where higher values correspond to stronger satiety/hunger)
Sleep quality and timing | 2 weeks (PSQI) and 14 days (ActiGraph, sleep diary)
  Sleep quality as assessed by the Pittsburgh Sleep Quality Index (PSQI score, which ranges from 0-21, where higher values correspond to worse sleep quality) and by the ActiGraph device; sleep timing (sleep onset and offset) as monitored using a sleep diary
Physical activity | 14 days
  24-h physical activity as monitored by an ActiGraph device
Expression of metabolic genes in adipose tissue | 2 weeks
  RNA-Seq analysis of subcutaneous adipose tissue samples
Social and economic decision behaviour | 2 weeks
  Assessed by computer tests together with the Barratt Impulsiveness Scale short version (BIS-15 with a score between 15 and 60, where higher values correspond to higher impulsiveness) and the UCLA Loneliness Scale (with a score between 20 and 100, where higher values correspond to higher subjectively perceived loneliness)

OTHER OUTCOMES:
Gene expression in peripheral mononuclear blood cells (PBMC) | 2 weeks
  mRNA expression of clock, metabolic and inflammatory genes
Internal circadian phase | 2 weeks
  Circadian phase as assessed using the BodyTime assay in isolated CD14+ blood monocytes

CONTACTS AND LOCATIONS:
Locations (1):
- German Institute of Human Nutrition Potsdam-Rehbruecke, Nuthetal, Germany

REFERENCES:
- [Derived] Peters B, Koppold-Liebscher DA, Schuppelius B, Steckhan N, Pfeiffer AFH, Kramer A, Michalsen A, Pivovarova-Ramich O. Effects of Early vs. Late Time-Restricted Eating on Cardiometabolic Health, Inflammation, and Sleep in Overweight and Obese Women: A Study Protocol for the ChronoFast Trial. Front Nutr. 2021 Nov 15;8:765543. doi: 10.3389/fnut.2021.765543. eCollection 2021. PMID 34869534